CLINICAL TRIAL: NCT06568042
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled, Dose-Finding Study Evaluating LY3848575 in Chronic Neuropathic Pain Associated With Distal Sensory Polyneuropathy
Brief Title: Effects of LY3848575 Versus Placebo in Participants With Painful Distal Sensory Polyneuropathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18825; J4F-MC-CYAB (Other: Eli Lilly and Company); 2024-513435-24-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Neuropathic Pain; Distal Sensory Polyneuropathy
Keywords: Peripheral Neuropathy; Diabetic Peripheral Neuropathy; Chemotherapy Induced Peripheral Neuropathy; HIV Induced Peripheral Neuropathy
MeSH Terms: conditions — Neuralgia; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3848575 Dose 1 (Experimental): LY3848575 low dose administered subcutaneously (SC).
  Interventions: Drug: LY3848575
- LY3848575 Dose 2 (Experimental): LY3848575 mid dose administered SC.
  Interventions: Drug: LY3848575
- LY3848575 Dose 3 (Experimental): LY3848575 high dose administered SC.
  Interventions: Drug: LY3848575
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3848575 — Administered SC
  Arms: LY3848575 Dose 1; LY3848575 Dose 2; LY3848575 Dose 3
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how safe and how well a treatment works compared to placebo for people with nerve pain that begins in their feet and moves up the leg to just below the knee.

Participation may last up to 30 weeks including screening.

ELIGIBILITY:
Inclusion Criteria:

* Have a Visual Analog Scale (VAS) pain value ≥40 and <95 at screening.
* Presence of painful distal sensory polyneuropathy (DSP) without prominent motor or autonomic features with gradual or insidious onset with a minimum duration of 6 months and a known cause of nerve injury, such as metabolic, toxic exposure, nutritional, immunologic, infectious, hereditary, multifactorial, or no known cause identified (idiopathic), of symmetrical nature and in lower extremities (with or without involvement of the hands).
* Are willing to maintain a consistent regimen of any ongoing nonpharmacologic pain- relieving therapies and/or nutritional supplements and will not start any new nonpharmacologic pain-relieving therapies and/or nutritional supplements during study participation.
* Are willing to discontinue all medications taken for chronic pain conditions, except the allowed pain medications.
* Individuals NOT of childbearing potential may participate in the trial. Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Other etiologies of pain that may not be due to DSP or confound the assessment due to painful DSP.
* Have had a procedure within the past 6 months intended to produce permanent sensory loss in the target area of interest.
* Have not achieved glycemic control on a stable diabetes treatment regimen for at least 90 days prior to screening, have a healthcare provider who manages the participants' diabetes, and have a hemoglobin A1c (HbA1c) >11% at screening.
* Cancer within 2 years of baseline, except for:

  * cutaneous basal cell or squamous cell carcinoma resolved by excision, or
  * cancer treatment which led to chemotherapy that caused distal sensory polyneuropathy.
* Are, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.
* Have a surgery planned during the study for any reason.
* History of chronic alcohol, illicit drug, or narcotic use disorder within 2 years prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Average Pain Intensity Numeric Rating Scale (API-NRS) | Baseline, Week 12

SECONDARY OUTCOMES:
Mean Change from Baseline in Worst Pain Intensity Numeric Rating Scale (WPI-NRS) | Baseline, Week 12
Mean Change from Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Custom Form (CF) v1.1 | Baseline, Week 12
Mean Change from Baseline in Pain Interference with Sleep | Baseline, Week 12
Mean Change from Baseline in PROMIS Short Form (SF) Physical Functioning (PF) 10a (PROMIS PF 10a) | Baseline, Week 12
Mean Change from Baseline in PROMIS (SF) Sleep Disturbance 8b (PROMIS SD 8b) | Baseline, Week 12
Mean Change from Baseline in 36-Item Short Form Health Survey Version 2 (SF-36 v2) | Baseline, Week 12
Mean Change from Baseline in Patient's Global Impression (PGI) of Illness Severity as Measured by PGI-Severity | Baseline, Week 12
Mean Overall Improvement as Measured by Patient's Global Impression of Change | Week 12
Use of Rescue Medication | Baseline up to Week 12
Pharmacokinetic (PK): Serum Concentration of LY3848575 | Baseline up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (76):
- United States (24):
  - MD First Research - Chandler, Chandler, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Accel Research Sites - St. Pete-Largo Clinical Research Unit, Largo, Florida
  - Design Neuroscience Center, Miami Lakes, Florida
  - Conquest Research - Orlando, Orlando, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Conquest Research, Winter Park, Florida
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Mid Hudson Medical Research, New Windsor, New York
  - University of Rochester Medical Center, Rochester, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - New Phase Research and Development, Knoxville, Tennessee
  - Cedar Health Research, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (7):
  - Med Trust Research, Courtice
  - Dawson Clinical Research Inc., Guelph
  - Premier Clinical Trial Network, Hamilton
  - OCT Research ULC, Kelowna
  - Genge Partners, Montreal
  - Richmond Clinical Trials, Richmond
  - Bluewater Clinical Research Group Inc., Sarnia
- Germany (5):
  - FutureMeds GmbH, Berlin
  - Studienzentrum Dr. Bischof GmbH, Böblingen
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - ZNS Siegen, Siegen
  - Studienzentrum Nord-West, Westerstede
- Japan (18):
  - St. Luke's International Hospital, Chūōku
  - Chugoku Central Hospital, Fukuyama-shi
  - Mito Medical Center, Higashiibaraki
  - Rinku General Medical Center, Izumisano
  - Sagara Hospital, Kagoshima
  - Kamezawa Clinic, Kasugai
  - The Cancer Institute Hospital of JFCR, Kōtō City
  - Kikuchi Naika Clinic, Maebashi
  - Aizawa Hospital, Matsumoto
  - Kojunkai Daido Hospital, Nagoya
  - Nishinomiya Municipal Central Hospital, Nishinomiya
  - Medical Corporation Sato Medical clinic, Ootaku
  - Minamiosaka Hospital, Osaka
  - Fujigaki Clinic, Ōita
  - Saga-Ken Medical Centre Koseikan, Saga
  - Asama General Hospital, Saku
  - Tokyo Shinagawa Hospital, Shinagawa-ku
  - Niwa Family Clinic, Tokyo
- Mexico (8):
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Investigación Clínica Cuernavaca, S.C., Cuernavaca
  - Centro de Investigación Clínica y Medicina Traslacional (CIMeT), Guadalajara
  - Health Pharma Querétaro, Juriquilla
  - Grupo Medico Camino Sc, Mexico City
  - Medical Care and Research SA de CV, Mérida
  - Cicmex Centro de Investigación Clínica de México, Morelia
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
- Poland (8):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Centrum Medyczne NEUROMED, Bydgoszcz
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk
  - Neuro-Care Sp. z o.o. sp. kom., Katowice
  - Diamond Clinic, Krakow
  - Santa Familia PTG Lodz, Lodz
  - Nzoz Neuro-Kard Ilkowski i Partnerzy SPL, Poznan
  - MICS Centrum Medyczne Warszawa - Chłodna, Warsaw
- South Korea (6):
  - Chosun University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Related Info — http://trials.lilly.com/en-US/trial/530315